CLINICAL TRIAL: NCT07231172
Title: Frequency of Post-stroke Fatigue and Its Relationship With Clinical Parameters
Brief Title: Post-stroke Fatigue and Clinical Parameters
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşe A Küçükdeveci, MD, Clinical Professor, Ankara University
Other Study IDs: İ07-516-24
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Fatigue; Poststroke Fatigue
Keywords: Fatigue, Stroke,; Frequency
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the frequency of post-stroke fatigue (PSF) in patients experiencing their first-ever stroke and admitted to our clinic. PSF is a common and debilitating condition that significantly impacts patients' recovery and quality of life. The study will also explore the association between fatigue severity and various demographic and clinical factors such as age, gender, stroke type and duration, pain, mood disorders, sleep quality, motor and cognitive functions, spasticity, physical capacity, ambulation, independence in daily living activities, and health-related quality of life. Patients over 18 years old, at least three months post-stroke, and meeting specific inclusion criteria will be recruited. Fatigue will be assessed using validated scales including the Fatigue Severity Scale and Visual Analog Scale-Fatigue. Additional assessments will measure pain, anxiety, depression, sleep disturbances, motor and cognitive status, spasticity, physical endurance, functional mobility, and daily activity independence. The findings are expected to contribute to a better understanding of PSF and help inform more effective rehabilitation strategies.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization, stroke is defined as "rapidly developing clinical manifestations of focal (or global) impairment of cerebral function that lasts longer than 24 hours or may result in death and has no apparent cause other than vascular origin". Stroke is the second leading cause of death in the world. It is also the leading cause of disability and accounts for a significant proportion of hospital admissions and health expenditures in industrialized societies. Stroke has many complications, one of which is fatigue. Fatigue can be defined as a decrease in physical and/or mental performance resulting from changes in central, psychological and/or environmental factors. Normal fatigue is a generalized state of tiredness resulting from overexertion and improves with rest. In contrast, "pathologic fatigue", often experienced by patients with neurological disorders, is chronic fatigue unrelated to previous levels of exertion and usually does not improve with rest. Post-stroke fatigue can be considered as a type of pathologic fatigue. Post-stroke fatigue is one of the most common symptoms 3 months after stroke. Half of the patients may still experience fatigue 1 year after stroke and this condition may last for years. The prevalence of post-stroke fatigue has been reported to vary between 39% and 68%. Post-stroke fatigue negatively affects the quality of life of stroke patients and constitutes a significant barrier to recovery, especially in participation in rehabilitation programs. Therefore, understanding post-stroke fatigue is an important issue for healthcare professionals in terms of implementing effective rehabilitation programs in patients with stroke. However, little is known about the etiology and effective management of post-stroke fatigue. Numerous factors have been shown to be associated with post-stroke fatigue, including age, gender, depression, stroke severity, stroke type and lesion location, pain, but these risk factors are not consistent across all studies. The lack of appropriate objective measurement tools may be one of the reasons for the poor understanding of post-stroke fatigue. Several tools are available to assess fatigue, including the Fatigue Rating Scale, Fatigue Impact Scale, Fatigue Severity Scale (FSS) and Visual Analogue Scale-Fatigue. The Fatigue Severity Scale (FSS) is the most commonly used fatigue assessment scale in stroke patients and was originally developed to measure fatigue in patients with Multiple Sclerosis and Systemic Lupus Erythematosus. In the literature, there are studies investigating the frequency of fatigue after stroke and its relationship with various demographic and clinical parameters. In our country, there are a few studies evaluating the frequency of fatigue after stroke. There is no complete clarity in terms of both the frequency and the factors associated with fatigue in the studies. Our primary aim in this study is to determine the frequency of post-stroke fatigue in first-time stroke patients admitted to our clinic. Our secondary aim is to evaluate the relationship between fatigue severity and demographic and clinical characteristics of the patients such as age, gender, education level, stroke type, stroke duration and severity of pain, anxiety, depression, sleep status, motor and cognitive function, spasticity, physical capacity, functional ambulation, level of independence in activities of daily living and health-related quality of life.

Method: The study will include patients who were diagnosed with stroke for the first time according to the World Health Organization definition, who were over 18 years of age, whose general condition was stable after stroke and at least 3 months have passed since the event, among the patients followed up in the Department of Physical Medicine and Rehabilitation of Ankara University Faculty of Medicine Ibn-i Sina and Cebeci hospitals. This study will be conducted within the scope of good clinical practices and all patients will be asked to give consent to the study by reviewing the informed consent form before the study.

Inclusion Criteria:

* Being diagnosed with stroke according to definition by the World Health Organization
* Being over 18 years of age
* Having had a stroke confirmed by Computed Tomography (CT) and/or Magnetic Resonance Imaging (MRI)
* At least 3 months after stroke
* At least stage 2 according to the Functional Ambulation Classification
* Agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* Previous history of stroke
* Communication problems due to reasons such as aphasia and dementia
* Patients who are illiterate
* Cognitive functional impairment who cannot take commands (MMSE<24)
* Dİagnoses such as cancer, heart failure, liver failure, renal failure that may cause fatigue
* Signs of systemic infection
* History of subarachnoid hemorrhage

Demographic information (gender, age, height, weight, body mass index, occupation), medical history, type of lesion (ischemic, hemorrhagic), duration of disease, laboratory values such as vitamin B12, vitamin D, hemoglobin and albumin levels and current treatments will be obtained from the patients who agree to participate in the study and meet the inclusion criteria and this information will be recorded in the patient follow-up form. Fatigue Severity Scale (FSS) will be used to assess fatigue after stroke. In addition, the Visual Analog Scale-Fatigue (VAS-Fatigue) will be used to determine the severity of fatigue. Pain severity will be assessed using the Visual Analog Scale-Pain (VAS-Pain), depression and anxiety will be assessed using the Hospital Anxiety and Depression Scale, sleep quality will be assessed using the Athens Insomnia Scale, motor function will be assessed using the Brunnstrom Motor Recovery Staging, and cognitive function will be assessed using the Mini Mental State Examination and Montreal Cognitive Assessment. The level of spasticity will be assessed with the Modified Ashworth Scale, physical capacity with the 6-minute walk test, functional ambulation with the Functional Ambulation Classification, independence in activities of daily living with the Modified Barthel Index, and health-related quality of life with the Stroke Impact Scale v3.0

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with stroke according to definition by the World Health Organization
* Being over 18 years of age
* Having had a stroke confirmed by Computed Tomography (CT) and/or Magnetic Resonance Imaging (MRI)
* At least 3 months after stroke
* At least stage 2 according to the Functional Ambulation Classification
* Agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* Previous history of stroke
* Communication problems due to reasons such as aphasia and dementia
* Patients who are illiterate
* Cognitive functional impairment who cannot take commands (MMSE<24)
* Dİagnoses such as cancer, heart failure, liver failure, renal failure that may cause fatigue
* Signs of systemic infection
* History of subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients admitted to Ankara University Faculty of Medicine, Physical Medicine and Rehabilitation Clinic
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Baseline
  The Fatigue Severity Scale was first used in 1989 by Krupp et al. to assess fatigue in patients with Multiple Sclerosis and Systemic Lupus Erythematosus. In stroke, a validity and reliability study was conducted for the first time by Nadarajah et al. in 2017. In our country, a validity and reliability study was conducted in stroke patients by Özyemişçi-Taşkıran et al. in 2019. The FSS is a self-report questionnaire that measures the impact and severity of fatigue in daily life. The FSS consists of 9 items about fatigue scored on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). The total score is the arithmetic mean of the 9 item scores. The lowest score is 9 points and the highest is 63 points. A total score of 36 points or an average score of 4 or more means that the fatigue is pathological fatigue. The higher the FSS score, the greater the impact of fatigue on daily life. Patients are assessed by asking questions according to their fatigue in the last week.
Visual Analog Scale-Fatigue | Baseline
  Visual Analog Scale-Fatigue (VAS-Fatigue): The Visual Analog Scale is a 10 cm horizontal line with a legend at each end and is commonly used to measure pain levels. The VAS has been modified and renamed VAS-F to measure pathologic fatigue in cancer. One end of the line (0) indicates no fatigue and the other end (10) indicates unbearable fatigue. The patient will be asked to mark the level of fatigue felt during the last 1 week on a 10 cm line. The possible score will be between 0 and 10, with a higher score indicating a high degree of fatigue.

SECONDARY OUTCOMES:
Visual Analog Scale-Pain | Baseline
  VAS-Pain is a 10 cm horizontal line on which the patient's pain intensity is evaluated. One end of the line (0) indicates no pain and the other end (10) indicates unbearable pain. The patient will be asked to mark on this 10 cm line the level of pain they have felt in their body in the last 1 week. The possible score will be between 0 and 10, with a higher score indicating a higher degree of pain.
Hospital Anxiety and Depression Scale | Baseline
  The HADS is a 14-item scale including 7 anxiety (HADS-A) and 7 depression (HADS-D) symptoms. The aim of the scale is not to make a diagnosis, but to identify the risk group by screening for anxiety and depression in patients with physical illness in a short time. Each item in the scale is evaluated with a four-point Likert scale scored between 0-3. The maximum total score of each subgroup is 21, and scores between 0-7 are considered normal, while scores of 11 and above are considered mood disorders.
Athens Insomnia Scale | Baseline
  AİS is a psychometric self-assessment tool developed by Soldatos et al. to determine the severity and impact of insomnia encountered in a wide variety of clinical and research settings. It consists of eight items: Sleep induction, awakenings during the night, final awakening earlier than desired, total sleep duration, overall sleep quality, sense of well-being during the day, functioning capacity during the day (physical and mental), and sleepiness during the day. Each item is scored between 0-3 points. The higher the score, the poorer the sleep quality.
Brunnstrom Motor Recovery Staging | Baseline
  It is used to evaluate hand, upper and lower extremity motor function of patients after stroke. It evaluates patients' synergy patterns, muscle tone and developmental stages of isolated movements. There are 3 main headings: upper extremity, hand and lower extremity and each is graded between 1-7 (1: no movement 7: normal motor function).
Mini Mental State Examination | Baseline
  It has been shown that it can be used as a cognitive screening test in patients with brain injury. Scoring in the Mini Mental State Examination is between 0-30. Scores between 24 and 30 are considered normal, while scores of 23 and below usually indicate cognitive impairment.
Montreal Cognitive Assessment | Baseline
  The MoCA was developed as a rapid screening test for mild cognitive impairment. It is a 30-point test assessing visual/spatial-executive functions, naming, memory, attention, language, abstract thinking, calculation, delayed recall and orientation. Higher scores indicate better cognitive status. A score of 21 or above is considered normal.
Modified Ashworth Scale | Baseline
  MAS is the most preferred scale to assess spasticity in the clinic. The scale, which was defined by Ashworth by scoring in 4 categories between 0-3, was modified by Bohannon and Smith in 1987 and a 1+ parameter was added to the scoring
6 Minute Walk Test | Baseline
  The 6-minute walk test will be used to assess physical capacity. In this test, participants walk for 6 minutes at the maximum possible walking speed for a distance of 30 meters, with marked areas every 3 meters, without running. Participants should be rested before the test. Heart rate, blood pressure and oxygen saturation are recorded before and after the test, as well as walking distance at the end of the test. In our study, we will only record walking distance. Walking distance is an indicator of functional capacity. In this test, which is a close assessment method to the submaximal exercise test, healthy people can walk an average of 400-700 meters. Although 6DYT is frequently used in the clinic to evaluate treatment response in cardiac and pulmonary diseases, it is also a meaningful scale for functional capacity in stroke patients.
Functional Ambulation Classification | Baseline
  The FAS is an assessment scale that shows the ambulation level of patients, whether they can walk or not, or if they can walk, how much help they need. This scale was developed by Holden et al. in 1984 on patients with walking difficulties due to neurological impairment, including stroke patients. It is graded from 0 to 5 (Grade 0 is non-ambulatory, Grade 5 is independent ambulation on all surfaces).
Modified Barthel Index | Baseline
  It is used to assess the level of independence in activities of daily living. It is an index that evaluates transfer, ambulation, use of wheelchair, climbing up and down stairs, feeding, dressing, personal care, bathing, toilet use, urinary and fecal continence parameters and evaluates patients in 5 groups according to these parameter scores. In these groups, which are evaluated from 1 to 5, 1 is considered as inadequate to do work, while 5 is considered as completely independent. The scale is evaluated over 100 points in total. A score of 100 indicates complete independence and a score of zero indicates complete dependence.
Stroke Impact Scale Version 3.0 | Baseline
  This multidimensional scale consists of 8 subsections (strength, hand function, activities of daily living, mobility, communication, emotion, memory and social participation) and a total of 59 questions. Each question scores the difficulty experienced in the past week on a 5-point Likert scale. A score of 1 indicates that the patient was unable to complete the item, while a score of 5 indicates that the patient completed the item without any difficulty. A low score indicates poor quality of life. In addition to the 8 subsections, the SİS v3.0 also assesses the perception of recovery after stroke with a 0-100 point visual analog scale (0: No recovery, 100: Complete recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe A. Küçükdeveci, Prof, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Duncan PW, Bode RK, Min Lai S, Perera S; Glycine Antagonist in Neuroprotection Americans Investigators. Rasch analysis of a new stroke-specific outcome scale: the Stroke Impact Scale. Arch Phys Med Rehabil. 2003 Jul;84(7):950-63. doi: 10.1016/s0003-9993(03)00035-2. PMID 12881816
- [Result] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Result] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723
- [Result] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Result] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Result] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Result] Macchiavelli A, Giffone A, Ferrarello F, Paci M. Reliability of the six-minute walk test in individuals with stroke: systematic review and meta-analysis. Neurol Sci. 2021 Jan;42(1):81-87. doi: 10.1007/s10072-020-04829-0. Epub 2020 Oct 16. PMID 33064231
- [Result] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Bour A, Rasquin S, Boreas A, Limburg M, Verhey F. How predictive is the MMSE for cognitive performance after stroke? J Neurol. 2010 Apr;257(4):630-7. doi: 10.1007/s00415-009-5387-9. Epub 2009 Nov 22. PMID 20361295
- [Result] Elhan AH, Kutlay S, Kucukdeveci AA, Cotuk C, Ozturk G, Tesio L, Tennant A. Psychometric properties of the Mini-Mental State Examination in patients with acquired brain injury in Turkey. J Rehabil Med. 2005 Sep;37(5):306-11. doi: 10.1080/16501970510037573. PMID 16203619
- [Result] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Brunnstrom S. Motor testing procedures in hemiplegia: based on sequential recovery stages. Phys Ther. 1966 Apr;46(4):357-75. doi: 10.1093/ptj/46.4.357. No abstract available. PMID 5907254
- [Result] Elbi H, Batum M, Ozturk EO, Balcan MV, Ak AK, Yilmaz H, Aydemir O. Adaptation into Turkish and Psychometric Properties of Athens Insomnia Scale. Noro Psikiyatr Ars. 2024 Apr 1;61(2):154-159. doi: 10.29399/npa.28575. eCollection 2024. PMID 38868854
- [Result] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. J Psychosom Res. 2000 Jun;48(6):555-60. doi: 10.1016/s0022-3999(00)00095-7. PMID 11033374
- [Result] Aben I, Verhey F, Lousberg R, Lodder J, Honig A. Validity of the beck depression inventory, hospital anxiety and depression scale, SCL-90, and hamilton depression rating scale as screening instruments for depression in stroke patients. Psychosomatics. 2002 Sep-Oct;43(5):386-93. doi: 10.1176/appi.psy.43.5.386. PMID 12297607
- [Result] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Result] Choi-Kwon S, Han SW, Kwon SU, Kim JS. Poststroke fatigue: characteristics and related factors. Cerebrovasc Dis. 2005;19(2):84-90. doi: 10.1159/000082784. Epub 2004 Dec 17. PMID 15608431
- [Result] Okuyama T, Akechi T, Kugaya A, Okamura H, Shima Y, Maruguchi M, Hosaka T, Uchitomi Y. Development and validation of the cancer fatigue scale: a brief, three-dimensional, self-rating scale for assessment of fatigue in cancer patients. J Pain Symptom Manage. 2000 Jan;19(1):5-14. doi: 10.1016/s0885-3924(99)00138-4. PMID 10687321
- [Result] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Result] Miller KK, Combs SA, Van Puymbroeck M, Altenburger PA, Kean J, Dierks TA, Schmid AA. Fatigue and pain: relationships with physical performance and patient beliefs after stroke. Top Stroke Rehabil. 2013 Jul-Aug;20(4):347-55. doi: 10.1310/tsr2004-347. PMID 23893834
- [Result] Ozyemisci-Taskiran O, Batur EB, Yuksel S, Cengiz M, Karatas GK. Validity and reliability of fatigue severity scale in stroke. Top Stroke Rehabil. 2019 Mar;26(2):122-127. doi: 10.1080/10749357.2018.1550957. Epub 2018 Nov 26. PMID 30475156
- [Result] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Result] Nadarajah M, Goh HT. Post-stroke fatigue: a review on prevalence, correlates, measurement, and management. Top Stroke Rehabil. 2015 Jun;22(3):208-20. doi: 10.1179/1074935714Z.0000000015. Epub 2015 Mar 17. PMID 25779764
- [Result] Hubacher M, Calabrese P, Bassetti C, Carota A, Stocklin M, Penner IK. Assessment of post-stroke fatigue: the fatigue scale for motor and cognitive functions. Eur Neurol. 2012;67(6):377-84. doi: 10.1159/000336736. Epub 2012 May 17. PMID 22614741
- [Result] Hinkle JL, Becker KJ, Kim JS, Choi-Kwon S, Saban KL, McNair N, Mead GE; American Heart Association Council on Cardiovascular and Stroke Nursing and Stroke Council. Poststroke Fatigue: Emerging Evidence and Approaches to Management: A Scientific Statement for Healthcare Professionals From the American Heart Association. Stroke. 2017 Jul;48(7):e159-e170. doi: 10.1161/STR.0000000000000132. Epub 2017 May 25. PMID 28546322
- [Result] Elbers RG, Rietberg MB, van Wegen EE, Verhoef J, Kramer SF, Terwee CB, Kwakkel G. Self-report fatigue questionnaires in multiple sclerosis, Parkinson's disease and stroke: a systematic review of measurement properties. Qual Life Res. 2012 Aug;21(6):925-44. doi: 10.1007/s11136-011-0009-2. Epub 2011 Oct 20. PMID 22012025
- [Result] Moos RH, Brennan PL, Schutte KK, Moos BS. Older adults' coping with negative life events: common processes of managing health, interpersonal, and financial/work stressors. Int J Aging Hum Dev. 2006;62(1):39-59. doi: 10.2190/ENLH-WAA2-AX8J-WRT1. PMID 16454482
- [Result] Blaauw E, Arensman E, Kraaij V, Winkel FW, Bout R. Traumatic life events and suicide risk among jail inmates: the influence of types of events, time period and significant others. J Trauma Stress. 2002 Feb;15(1):9-16. doi: 10.1023/A:1014323009493. PMID 11936726
- [Result] Tang WK, Chen YK, Liang HJ, Chu WC, Mok VC, Ungvari GS, Wong KS. Subcortical white matter infarcts predict 1-year outcome of fatigue in stroke. BMC Neurol. 2014 Dec 12;14:234. doi: 10.1186/s12883-014-0234-8. PMID 25496671
- [Result] Nadarajah M, Mazlan M, Abdul-Latif L, Goh HT. Test-retest reliability, internal consistency and concurrent validity of Fatigue Severity Scale in measuring post-stroke fatigue. Eur J Phys Rehabil Med. 2017 Oct;53(5):703-709. doi: 10.23736/S1973-9087.16.04388-4. Epub 2016 Oct 21. PMID 27768012
- [Result] Barker-Collo S, Feigin VL, Dudley M. Post stroke fatigue--where is the evidence to guide practice? N Z Med J. 2007 Oct 26;120(1264):U2780. PMID 17972987
- [Result] Chestnut TJ. Fatigue in stroke rehabilitation patients: a pilot study. Physiother Res Int. 2011 Sep;16(3):151-8. doi: 10.1002/pri.476. Epub 2010 May 18. PMID 24737613
- [Result] Gordon NF, Gulanick M, Costa F, Fletcher G, Franklin BA, Roth EJ, Shephard T; American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Physical activity and exercise recommendations for stroke survivors: an American Heart Association scientific statement from the Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Circulation. 2004 Apr 27;109(16):2031-41. doi: 10.1161/01.CIR.0000126280.65777.A4. No abstract available. PMID 15117863
- [Result] Schepers VP, Visser-Meily AM, Ketelaar M, Lindeman E. Poststroke fatigue: course and its relation to personal and stroke-related factors. Arch Phys Med Rehabil. 2006 Feb;87(2):184-8. doi: 10.1016/j.apmr.2005.10.005. PMID 16442970
- [Result] van der Werf SP, van den Broek HL, Anten HW, Bleijenberg G. Experience of severe fatigue long after stroke and its relation to depressive symptoms and disease characteristics. Eur Neurol. 2001;45(1):28-33. doi: 10.1159/000052085. PMID 11150837
- [Result] Skaner Y, Nilsson GH, Sundquist K, Hassler E, Krakau I. Self-rated health, symptoms of depression and general symptoms at 3 and 12 months after a first-ever stroke: a municipality-based study in Sweden. BMC Fam Pract. 2007 Oct 17;8:61. doi: 10.1186/1471-2296-8-61. PMID 17941995
- [Result] Kirkevold M, Christensen D, Andersen G, Johansen SP, Harder I. Fatigue after stroke: manifestations and strategies. Disabil Rehabil. 2012;34(8):665-70. doi: 10.3109/09638288.2011.615373. Epub 2011 Oct 13. PMID 21995298
- [Result] Staub F, Bogousslavsky J. Post-stroke depression or fatigue. Eur Neurol. 2001;45(1):3-5. doi: 10.1159/000052081. No abstract available. PMID 11205620
- [Result] De Groot MH, Phillips SJ, Eskes GA. Fatigue associated with stroke and other neurologic conditions: Implications for stroke rehabilitation. Arch Phys Med Rehabil. 2003 Nov;84(11):1714-20. doi: 10.1053/s0003-9993(03)00346-0. PMID 14639575
- [Result] Staub F, Bogousslavsky J. Fatigue after stroke: a major but neglected issue. Cerebrovasc Dis. 2001 Aug;12(2):75-81. doi: 10.1159/000047685. PMID 11490100
- [Result] Acciarresi M, Bogousslavsky J, Paciaroni M. Post-stroke fatigue: epidemiology, clinical characteristics and treatment. Eur Neurol. 2014;72(5-6):255-61. doi: 10.1159/000363763. Epub 2014 Sep 24. PMID 25277765
- [Result] Cumming TB, Packer M, Kramer SF, English C. The prevalence of fatigue after stroke: A systematic review and meta-analysis. Int J Stroke. 2016 Dec;11(9):968-977. doi: 10.1177/1747493016669861. Epub 2016 Oct 4. PMID 27703065
- [Result] Stroke--1989. Recommendations on stroke prevention, diagnosis, and therapy. Report of the WHO Task Force on Stroke and other Cerebrovascular Disorders. Stroke. 1989 Oct;20(10):1407-31. doi: 10.1161/01.str.20.10.1407. No abstract available. PMID 2799873
- [Result] Aho K, Harmsen P, Hatano S, Marquardsen J, Smirnov VE, Strasser T. Cerebrovascular disease in the community: results of a WHO collaborative study. Bull World Health Organ. 1980;58(1):113-30. PMID 6966542
- See also: Related Info — https://www.ftrdergisi.com/abstract.php?lang=tr&id=3208
- See also: Related Info — https://tjcvd.org/jvi.aspx?un=TBDHD-04834&volume=14&issue=3
- See also: Related Info — https://www.jpmrs.org/uploads/973440954215479.pdf
- See also: Related Info — https://www.researchgate.net/publication/301778685_Hastane_Anksiyete_ve_Depresyon_Olcegi_Turkce_Formunun_Gecerlilik_ve_Guvenilirlik_Calismasi_Reliability_and_Validity_of_the_Turkish_version_of_Hospital_Anxiety_and_Depression_Scale
- See also: Related Info — https://search.trdizin.gov.tr/tr/yayin/detay/105939
- See also: Related Info — https://www.ftrdergisi.com/uploads/sayilar/286/buyuk/106-116.pdf